CLINICAL TRIAL: NCT06234644
Title: Effects on Maze Activities on Mobility in Children With Down's Syndrome
Brief Title: Effects of Maze Activities in Down's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0747
Record Dates: First submitted 2023-12-26; First posted 2024-01-31 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
Keywords: Down's Syndrome; Mobility; Standardized Walking obstacle course (SWOC).
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): The Group A (experimental group) will receive the treatment with Standardized walking obstacle course (SWOC).
  Interventions: Other: Standardized Walking Obstacle Course (SWOC)
- Group B (Active Comparator): The Group B (Control group) will receive the treatment with conventional Gait training.
  Interventions: Other: Conventional Gait Training

INTERVENTIONS:
Other: Standardized Walking Obstacle Course (SWOC) — The Standardized Walking Obstacle Course (SWOC) is a test that allows interaction of a child with environmental demands and obstructions while examining differences in functional ambulation performances. The Group A (experimental group) will receive the treatment with Standardized walking obstacle course (SWOC), the group of 13 participants will receive the treatment. This group will receive therapy session for 45 min, thrice a week for 6 weeks, total sessions will be 18. 45 minutes session time will be divided into 15 min warm up period, 25 minutes of SWOC training and 5 minutes of cool down period.
  Arms: Group A
Other: Conventional Gait Training — Conventional gait training protocol including walking on a treadmill, parallel bar walk, seated marching. The Group B (Control group) will receive the treatment with conventional Gait training, the group of 13 participants will receive the treatment. This group will receive therapy session for 45 min, thrice a week for 6 weeks, total sessions will be 18. 45 minutes session time will be divided into 15 min warm up period, 25 minutes of Conventional gait training and 5 minutes of cool down period.
  Arms: Group B

SUMMARY:
Down's Syndrome is due to the chromosomal disorder in 47 chromosomes instead of 46, socalled as Trisomy 21. The syndrome has several clinical symptoms including Cardiovascular,neurological, orthopedic, hormonal, cognitive and visual perceptual impairments. These childrenhave Developmental Delay. Children have hypermobility of joints, hypotonicity or ligamentous laxity, light to moderate obesity, due to underdeveloped respiratory and cardiovascular systemandshortstaturewhichleadtodecreaseinfunctionalambulation.Due to the low level of physical fitness, theseindividuals shows limitation in performing the functional tasks of daily living. The fundamental motor skill is Walking that facilitates the child to interact with the environment and helps indeveloping, social, motor and cognitive skills. Due to their delayed milestones and due to the irintellectual disability, environmental exposure is limited which hampers this fundamental skill.Hence it is necessary to asses the functional ambulation in these children.

This is a Randomized Controlled Trial that will be conducted in Rising Sun Institute Of Special Children. 26 participants will be allocated randomly into 2 groups Group A will receive the conventional interventions of Down's Syndrome but the group B will receive the mobility training with Standardized Walking Obstacle Course (SWOC). Tool used for this research will be a Standardized Walking Obstacle Course (SWOC) (that is used to measure stability and speed during gait in terms of time, number of steps, number of stumbles and number of steps off the path for each participant) and Timed up and go test (Valid for the functional mobility assessment of the children with DS). The data will be analyzed by SPSS version 21

DETAILED DESCRIPTION:
This study will be a randomized control trail used to compare the Effects of Maze Activities on Mobility in Children With Down's Syndrome. Subjects with Down's syndrome meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique. Assessment will be done by using time up and go test and Standardized Walking Obstacle Course (SWOC). Subjects in group A will receive the conventional intervention of gait training and Group B will receive the training on Standardized walking obstacle course.

ELIGIBILITY:
Inclusion Criteria:

* •Age 6 to 12 years of downs's syndrome children

  * Ambulatory Child who can walk without any assistive device(6)
  * Should follow commands and can perform 30 sec walk test.(6)

Exclusion Criteria:

* •Any congenital Cardiac Anomaly

  * Visual and Hearing Deficits
  * Any surgical intervention for the last 6 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Timed up and Go Test (TUG) | 6 weeks
  Time up and go test is used to assess the balance and stability of a children with different abilities. It involves timing how long it takes for a child to stand up from a chair, walk a short distance, turn around, walk back, and sit down while turning 180 degree.
  Interpretation: < 10 seconds = normal, < 20 seconds = good mobility, can go out alone, mobile without a gait aid. < 30 seconds = problems, cannot go outside alone, requires a gait aid. A score of more than or equal to fourteen seconds has been shown to indicate high risk of falls.
Standardized Walking Obstacle Course (SWOC) | 6 weeks
  It is used to measure stability and speed during gait in terms of time, number of steps, number of stumbles and number of steps off the path.Standardized walking obstacle course (SWOC) It is used to measure stability and speed during gait in terms of time, No of steps, No of stumbles, No of step off the path It is used to measure stability and speed during gait in terms of time, number of steps, number of stumbles and number of steps off the path. It was assessed under three conditions such as walk with arms free, walk with tray and walk with sunglasses.

CONTACTS AND LOCATIONS:
Overall Officials: Fibha Tariq, MS*, Principal Investigator — Riphah international university lahore
Locations (1):
- Riphah international university lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kott KM, Held S, Franjoine MR. Reference data for performances on the standardized walking obstacle course in children developing typically. Gait Posture. 2016 Sep;49:398-401. doi: 10.1016/j.gaitpost.2016.08.001. Epub 2016 Aug 2. PMID 27505143